CLINICAL TRIAL: NCT04881565
Title: Losing Balance to Prevent Falls After Spinal Cord Injury
Brief Title: Losing Balance to Prevent Falls After Spinal Cord Injury (RBT+FES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-5210
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries
Keywords: balance training; falls
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The clinical measures of balance, strength and proprioception will be administered by a physical therapist blind to group allocation. The physical therapist will not work at the facility where the research is being conducted, therefore reducing the likelihood of a breach of allocation concealment. If a breach occurs, it will be reported in the final publication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reactive balance training plus functional electrical stimulation (Experimental)
  Interventions: Other: Reactive balance training
- Reactive balance training (Active Comparator)
  Interventions: Other: Reactive balance training

INTERVENTIONS:
Other: Reactive balance training — During each one-hour session, participants will experience 40-50 perturbations (i.e. approximately one perturbation per training minute) during standing and/or walking activities. The perturbations will be applied in any direction (e.g. forwards, sideways, backwards, etc.) To create a perturbation, the researcher will apply unexpected pushes or pulls to a safety harness at waist level. The perturbation will be sufficient in magnitude to elicit a stepping response from the participant. Throughout the session, participants will complete challenging balance tasks, customized to their ability level. Balance tasks will be organized into five categories: stable, quasi-mobile, mobile, unpredictable and participant-selected.

SUMMARY:
Falls are a health crisis that cost health care systems billions of dollars/year. This crisis is especially relevant for individuals living with incomplete spinal cord injury (iSCI); 78% fall at least once annually. In able-bodied individuals, falls are prevented by taking reactive steps; however, these reactions are impaired after iSCI. Research in stroke and geriatric rehabilitation showed that reactive balance training (RBT), which targets reactive stepping, prevents falls. We developed a modified version of RBT for the iSCI population. RBT resulted in fewer falls post-training compared to dose-matched, conventional balance training. However, only those who were able to take a step independently and without upper limb support were able to participate in RBT, limiting the applicability of this promising fall prevention method. To address this limitation, we will integrate functional electrical stimulation into RBT (RBT+FES). Our study aims to provide a preliminary evaluation of the efficacy of RBT+FES in participants with chronic, motor iSCI. We will complete a pilot randomized clinical trial (RCT) with 22 participants with iSCI. Participants will be randomly allocated to RBT+FES or to RBT alone (i.e. without FES). They will complete 18 training sessions over 6 weeks (3 sessions/week). Clinical and biomechanical assessments of balance, strength and proprioception will be completed before training, immediately after training, and six months post-training. Falls will be monitored for six months after training through an online survey and regular phone calls. Performance on clinical and biomechanical measures and fall data will be compared between groups. This research will inform the need for, and design of, a larger RCT, and has the potential to transform fall prevention after iSCI.

ELIGIBILITY:
Inclusion Criteria:

1. Participant sustained a traumatic or non-progressive, non-traumatic motor iSCI (i.e. AIS C or D).
2. Injury occurred more than a year prior to study enrollment (when natural recovery has plateaued).8,9
3. Participant is ≥18 years old.
4. Participant can attend three training sessions/week for six weeks (i.e. has reliable transportation).
5. Participant is able to stand for >30 seconds without upper limb support or assistance (i.e. scores 2/4 on item two of the Berg Balance Scale, Standing Unsupported10). This criterion ensures the participant will be able to participate in upright balance exercises.
6. Participant requires physical assistance, a gait aid or a brace to ambulate 10 meters (i.e. self-selected score of 1-19 on the Walking Index for Spinal Cord Injury (WISCI) II).

Exclusion Criteria:

1. Participant presents with contraindications to FES (i.e. implanted electronic device, radiation in past six months, active deep vein thrombosis, pregnancy).12
2. Participant presents with other conditions besides iSCI that affect balance (e.g. vestibular disorder, brain injury).
3. Participant has a pressure injury (>grade 2) on the pelvis or trunk where the safety harness will be applied, or on the foot where the foot switch will be applied.
4. Participant has a history of a lower limb fragility fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Change from baseline to 6-month follow-up
mini-Balance Evaluation Systems Test | Change from baseline to 6-month follow-up
Activities-specific Balance Confidence Scale | Change from baseline to 6-month follow-up
Falls Efficacy Scale - International | Change from baseline to 6-month follow-up
Isometric strength | Change from baseline to 6-month follow-up
  The isometric strength of eight lower extremity muscle groups (hip extensors, hip flexors, hip abductors, hip adductors, knee extensors, knee flexors, ankle plantarflexors, ankle dorsiflexors) will be tested bilaterally using hand-held dynamometry.
Proprioception of the ankle joints | Change from baseline to 6-month follow-up
  To test proprioception, participants will assume a supine position with their eyes closed while the blinded assessor moves the ankle joint six times slowly through 10° of dorsiflexion (i.e. up) or plantarflexion (i.e. down). Participants will be asked to state the perceived direction of movement (i.e. up or down). This process will be repeated six times for each ankle, with a score of 1 assigned for each correct response. Each ankle will receive a maximum score of 6 for a total possible score of 12 (i.e. 2 joints x 6 trials/joint).
Lean-and-Release Test | Change from baseline to 6-month follow-up
  A lab-based assessment of reactive stepping ability (with and without FES).
Tracking falls | Change from beginning to end of 6-month follow-up period
  Falls will be monitored for six months following the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kristin E Musselman, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- KITE-Toronto Rehabilitation Institute, UHN, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No